CLINICAL TRIAL: NCT03358966
Title: Energy Expenditure in Chronic Kidney Disease: a Doubly Labelled Water Study
Brief Title: Energy Expenditure in Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Collaborators: University of Hertfordshire (Other)
Responsible Party: Sponsor
Other Study IDs: 08/H/0311/103 (REC No.); RP27/2010 (Other Grant/Funding Number: Kidney Research UK)
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-10

CONDITIONS: Kidney Diseases; Chronic Kidney Diseases
Keywords: chronic kidney disease; energy expenditure; metabolic rate
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early to moderate CKD (stage 1-3): 40 patients with CKD stage 1-3. All subjects performed a comprehensive metabolic analysis including measurement of Resting Energy Expenditure using indirect calorimetry, bioimpedance, doubly-labelled water technique and body size measures. Physical activity was assessed using a Stanford 7 day recall questionnaire.
  Interventions: Other: Doubly-labelled water technique; Other: Resting Energy Expenditure
- Advanced CKD (stage 4-5): 40 patients with CKD stage 4-5. All subjects performed a comprehensive metabolic analysis including measurement of Resting Energy Expenditure using indirect calorimetry, bioimpedance, doubly-labelled water technique and body size measures. Physical activity was assessed using a Stanford 7 day recall questionnaire.
  Interventions: Other: Doubly-labelled water technique; Other: Resting Energy Expenditure

INTERVENTIONS:
Other: Doubly-labelled water technique
Other: Resting Energy Expenditure — Resting energy expenditure represents the amount of calories required for a 24-hour period by the body during a non-active period.

SUMMARY:
Patients with kidney disease need accurate advice on their diet. Researchers know very little about energy needs and nutritional requirements in kidney patients. Simple tools are needed to calculate calorie requirements so that good bed-side advice can be given to patients, and to allow cost-effective research. This study aimed to measur energy requirements in kidney disease using a gold-standard safe and very accurate method called the "doubly labelled water technique". The study has compared measurements with less costly measurements obtained using a device which measures oxygen content of air breathed out. The study has also measured physical activity levels with questionnaires.

DETAILED DESCRIPTION:
Background The function of the kidneys is to remove waste products of metabolism, and despite advances in treatment of CKD little is known about metabolic rate in renal disease. Increased knowledge about metabolic rate would have numerous potential benefits.

Little is known of the effects of metabolic rate on kidney disease. This study was designed to define the relationship of metabolic rate with degree of kidney function.

Study design and methods In an observational cohort study, the investigators studied Total Energy Expenditure in 80 patients with CKD stage 1-5 using the doubly-labelled water technique over a 14 day period. The group was divided such that half had stage 1-3 CKD and half stage 4-5. All subjects performed a comprehensive metabolic analysis including measurement of Resting Energy Expenditure using indirect calorimetry, bioimpedance, and body size measures. Physical activity was assessed using a Stanford 7 day recall questionnaire.

Data Analysis The data analysed will include determining the relationship between level of kidney disease as measured by eGFR and energy expenditure measured as Resting Energy Expenditure and doubly-labelled water Total Energy Expenditure. This will be determined by regression analysis. Additionally, comparison will be made between subjects with early-moderate (CKD stage 1-3) and advanced (CKD stage 4-5) CKD.

ELIGIBILITY:
Inclusion Criteria:

1. CKD stages 1-5 according to the MDRD equation eGFR
2. Age >18

Exclusion Criteria:

1. Abnormal thyroid stimulating hormone level or previous thyroid disorder
2. Active malignancy
3. Pregnancy
4. Intercurrent illness or infection
5. Hospital admission in month prior to enrolment
6. Surgery in 4 weeks prior to enrolment
7. HIV, Hepatitis B, Hepatitis C positive status
8. Tuberculosis in the 12 months prior to enrolment.
9. Active vasculitis or connective tissue disorder
10. Organ transplantation.
11. Treatment with immunosuppression, except low dose corticosteroids (<10mg/day prednisolone).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease who attended the renal clinics of the East and North Herts NHS Trust
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2008-09-01 (Actual); Primary Completion 2014-05-30 (Actual); Study Completion 2015-05-30 (Actual)

PRIMARY OUTCOMES:
Energy expenditure using doubly labelled water | 14 days

SECONDARY OUTCOMES:
Whole body bioimpedance | 1 day
Resting Energy Expenditure using indirect calorimetry | 1 day
Stanford 7 day recall questionnaire physical activity level | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Professor Ken Farrington, Study Chair — East and North Hertfordshire NHS Trust

IPD SHARING:
Plan to Share IPD: No